CLINICAL TRIAL: NCT06553326
Title: EndoStyle: Survey of Physicians on Endoscopic Image Style Transfer.
Brief Title: EndoStyle: Artificial Intelligence Image Transformation Tool for Colonoscopy
Acronym: EndoStyle
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AI05
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer; Colon Rectal Cancer
Keywords: colonoscopy; Artificial intelligence
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Positive control: The image shown to the participant belongs to the same colonoscopy shown in the 10 second video-sequence.
- Negative control: The image shown to the participant belongs to the same colonoscopy shown in the 10 second video-sequence.
- EndoStyle (intervention group): The image shown to the participant does not belong to the 10 second colonoscopy video-sequence but has been transformed with AI to simulate the style of the video.
  Interventions: Device: EndoStyle

INTERVENTIONS:
Device: EndoStyle — The EndoStyle system is able to transform the style of the different video-processor images.
  Groups: EndoStyle (intervention group)

SUMMARY:
The study addresses the limitations of current AI systems in gastrointestinal endoscopy, which are tipically trained with data from a single type of endoscopy processor and have limited expert-annotated images. The investigators aim to develop and validate EndoStyle, an AI system that can generate images in the style of various processors from a single reference image. EndoStyle will be tested by showing endoscopists colonoscopy sequences with different image types to determine if they can distinguish AI-transformed images. Success would enhance AI training for diverse clinical setups.

DETAILED DESCRIPTION:
The use of artificial intelligence (AI) in gastrointestinal endoscopy has become widespread. However, these systems are often only trained with data from a single type of endoscopy processor, which limits their applicability. In addition, the availability of images annotated by experts is limited, which affects data variability and thus the performance of AI systems.

The aim of this study is to develop a new artificial intelligence (AI) based system (EndoStyle) and validate its authenticity by means of a survey among physicians, which is able to generate multiple images in the style of different processor types (including Olympus, Pentax and Storz) from a single endoscopy reference image.

The investigators hypothesis is that the AI system is able to successfully change the image style of video processors, with the differences being imperceptible to the endoscopist's eye.

The methodology consists of showing to multiple endoscopists 28 colonoscopy sequences of 10 seconds duration each. In each one of them 3 images will be shown that can be all the possible combinations of images belonging to positive control, negative control, and Endostyle (intervention group). By performing a statistical comparison of the percentages of selected images for each group the investigators will be able to establish whether the participants are able to distinguish the images transformed by the AI.

If the results corroborate our hypothesis, our system could generate images that would allow a more customized training of AI systems for each clinical setup.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with experience in colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants to the survey will be physicians with experience in colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Perceptual Indistinguishability of AI-Transformed Endoscopic Images | 5 months
  Comparison of the accuracy for each study group.

SECONDARY OUTCOMES:
Time Taken for Image Identification | 5 months
  Time taken to assess the different tasks according to each study group.
Influence of regularly used processor | 5 months
  Influence of regularly used endscopy processor during clinical work for the perceptual indistinguishability of AI-transformed endoscopic images with defined processor classes
Influence of endoscopy experience | 5 months
  Influence of experience in endoscopy measured in lifetime performed colonscopies on perceptual indistinguishability of AI-transformed endoscopic images

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hann, MD, Principal Investigator — University Hospital of Würzburg
Locations (1):
- University Clinic of Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided